CLINICAL TRIAL: NCT04580641
Title: Allodynia and Sensorial Hypersensitivity in Patients With Migraine: Validation of a Specific Questionnaire
Brief Title: Validation of a Questionnaire for Allodynia in Migraine.
Acronym: Q-MIGAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2018 MOISSET (Q-MIGAL)
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Migraine
Keywords: migraine; allodynia; photophobia; phonophobia; osmophobia; central sensitization
MeSH Terms: conditions — Migraine Disorders; Hyperalgesia; Photophobia; Hyperacusis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with migraine: No medical intervention. All included subjects will filled in the questionnaire concerning migraine characteristics and associated symptoms.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A self-administered questionnaire will be completed by each study subject

SUMMARY:
Migraine is very frequent (15% of the general population). During attacks, many subjects with migraine have allodynia (pain induced by normally non-painful stimuli), photophobia (hypersensitivity to light), phonophobia (hypersensitivity to sound) or osmophobia (hypersensitivity to odours). The goal of the present study is to validate a new questionnaire made of 4 parts evaluating the presence of these 4 types of hypersensitivity, both during or between migraine attacks. It will allow to look for associations of these 4 symptoms and association of hypersensitivity with patients' or migraine's characteristics.

DETAILED DESCRIPTION:
The prevalence of migraine is around 15% worldwide (GBD 2016, Lancet Neurol 2018). During attacks, and even between attacks, especially when migraine frequency is high, many subjects with migraine present with photophobia, phonophobia, osmophobia or allodynia. These symptoms are though to correspond to central sensitization and can be found in animal models of migraine (Boyer et al., Pain 2017; Dallel et al., Cephalalgia 2018).

These 4 symptoms have been studied separately in previous studies but to date, there is no overall questionnaire evaluating these 4 sub-types of hypersensitivity. The investigators have constituted a questionnaire based on previous validated questionnaires that have been translated into French (Lipton et al., 2008 for cutaneous allodynia; Choi et al., 2009 for photophobia), a previous questionnaire validated in French (Khalfa et al, 2002 for phonophobia) and created a few questions for each of the 4 symptoms, including osmophobia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fulfilling 2018 international headache society criteria for migraine.
* Age > 17 years.
* Written consent.

Exclusion Criteria:

* Presence of neurological comorbidities that could lead to sensorial or sensitive abnormalities
* Presence of dermatological comorbidities that could lead to sensorial or sensitive abnormalities
* Presence of ENT comorbidities that could lead to sensorial or sensitive abnormalities
* Significant cognitive dysfunction precluding proper completion of the self-administered questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects fulfilling 2018 international headache society criteria for migraine
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Predictive factors of allodynia/hypersensitivity in subjects with migraine | baseline
  Correlations between scores on specific questionnaires evaluating allodynia/hypersensitivity (cutaneous allodynia with the questionnaire by Lipton et al., 2008, osmophobia with a home-made questionnaire rated from 0 to 4, photophobia with the questionnaire by Choi et al., 2009, phonophobia with the questionnaire by Khalfa et al., 2002), patients characteristics (age, sex, Body mass index, habits, score on the Hospital Anxiety and Depression scale) and migraine characteristics (presence of aura or not, migraine duration in years, migraine frequency in attacks per month, pain intensity during migraine attacks rated from 0 to 4).

SECONDARY OUTCOMES:
Predictive factors of cutaneous allodynia in subjects with migraine | baseline
  Correlations between score on the 12-item Allodynia Symptom Checklist (Lipton et al., 2008) (score from 0 to 24 with higher values indicating higher level of allodynia), patients characteristics (age in years, sex, body mass index in kg/m², consumption of alcohol and tobacco, score on the Hospital Anxiety and Depression scale) and migraine characteristics (presence of aura or not, migraine duration in years, migraine frequency in attacks per month, pain intensity during migraine attacks rated from 0 to 4) .
Predictive factors of photophobia in subjects with migraine | baseline
  Correlations between scores on two specific questionnaires evaluating photophobia (Choi et al., 2009; binary score for presence or absence of photophobia and home-made questionnaire with score from 0 to 4 with higher values indicating higher level of phonophobia), patients characteristics (age in years, sex, body mass index in kg/m², consumption of alcohol and tobacco, score on the Hospital Anxiety and Depression scale) and migraine characteristics (presence of aura or not, migraine duration in years, migraine frequency in attacks per month, pain intensity during migraine attacks rated from 0 to 4).
Predictive factors of phonophobia in subjects with migraine | baseline
  Correlations between scores on a questionnaire evaluating phonophobia (Khalfa et al. 2002, score from 0 to 42 with higher values indicating higher level of phonophobia), patients characteristics (age in years, sex, body mass index in kg/m², consumption of alcohol and tobacco, score on the Hospital Anxiety and Depression scale) and migraine characteristics, (presence of aura or not, migraine duration in years, migraine frequency in attacks per month, pain intensity during migraine attacks rated from 0 to 4).
Predictive factors of osmophobia in subjects with migraine | baseline
  Correlations between scores on a specific home-made questionnaire evaluating osmophobia (score from 0 to 4 with higher values indicating higher level of osmophobia), patients characteristics (age in years, sex, body mass index in kg/m², consumption of alcohol and tobacco, score on the Hospital Anxiety and Depression scale) and migraine characteristics (presence of aura or not, migraine duration in years, migraine frequency in attacks per month, pain intensity during migraine attacks rated from 0 to 4).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Moisset, MD, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (14):
- France (14):
  - CH d'Annecy, Centre d'Etude et de Traitement de la Douleur, Annecy
  - Cabinet de Neurologie, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Centre d'Etude et de Traitement de la Douleur, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Service de Neurologie, Clermont-Ferrand
  - CH Emile Roux Le Puy en Velay, Service de Neurologie, Le Puy-en-Velay
  - CHU de Lille, Service de Neurologie, Lille
  - CHU de Lyon, Hôpital Pierre Wertheimer, Service de neurologie fonctionelle et épileptologie, Lyon
  - Assistance Publique - Hôpitaux de Marseille, CHU La Timone, Centre d'Evaluation et Traitement de la Douleur, Marseille
  - CHU de Montpellier, Service de Neurologie, Montpellier
  - CHU de Nantes, Service de Neurologie, Nantes
  - CHU de Nice, Département Evaluation et Traitement de la Douleur, Nice
  - Assistance Publique - Hôpitaux de Paris, CHU Lariboisière, Service de Neurologie, Paris
  - CHU de Rouen, Service de Neurologie, Rouen
  - CH de Vichy, Service de Neurologie, Vichy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi JY, Oh K, Kim BJ, Chung CS, Koh SB, Park KW. Usefulness of a photophobia questionnaire in patients with migraine. Cephalalgia. 2009 Sep;29(9):953-9. doi: 10.1111/j.1468-2982.2008.01822.x. Epub 2009 Feb 27. PMID 19298545
- [Background] Lipton RB, Bigal ME, Ashina S, Burstein R, Silberstein S, Reed ML, Serrano D, Stewart WF; American Migraine Prevalence Prevention Advisory Group. Cutaneous allodynia in the migraine population. Ann Neurol. 2008 Feb;63(2):148-58. doi: 10.1002/ana.21211. PMID 18059010
- [Background] Khalfa S, Dubal S, Veuillet E, Perez-Diaz F, Jouvent R, Collet L. Psychometric normalization of a hyperacusis questionnaire. ORL J Otorhinolaryngol Relat Spec. 2002 Nov-Dec;64(6):436-42. doi: 10.1159/000067570. PMID 12499770